CLINICAL TRIAL: NCT03064295
Title: Whole-Heart Myocardial Blood Flow Quantification Using Magnetic Resonance Imaging
Brief Title: Whole-Heart Myocardial Blood Flow Quantification Using MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Debiao Li, PhD, Director, Biomedical Imaging Research Institute, Cedars-Sinai Medical Center
Other Study IDs: 42972; 1R01HL124649 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Coronary Microvascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Microvascular Angina | interventions — Myocardial Perfusion Imaging; Magnetic Resonance Imaging; Contrast Media; gadobutrol; gadobenic acid; regadenoson; Adenosine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Healthy Volunteers: 60 healthy male or female (18 or older) adults will receive Myocardial Perfusion Cardiac MRI, including administration of contrast and a pharmacologic stress agent
  Interventions: Device: Myocardial Perfusion Cardiac MRI.; Drug: Contrast; Drug: Pharmacologic Stress Agent
- CAD Patients: 110 male or female adults (18 or older) who have undergone clinical myocardial perfusion imaging at CSMC and been diagnosed with Coronary Disease (CAD) will receive Myocardial Perfusion Cardiac MRI, including administration of contrast and a pharmacologic stress agent.
  Interventions: Device: Myocardial Perfusion Cardiac MRI.; Drug: Contrast; Drug: Pharmacologic Stress Agent
- CMD Patients: 50 female adults (21 or older) who have undergone coronary reactivity testing at CSMC and been diagnosed with coronary microvascular disease (CMD) will receive Myocardial Perfusion Cardiac MRI, including administration of contrast and a pharmacologic stress agent.
  Interventions: Device: Myocardial Perfusion Cardiac MRI.; Drug: Contrast; Drug: Pharmacologic Stress Agent

INTERVENTIONS:
Device: Myocardial Perfusion Cardiac MRI. — MRI with administration of a contrast drug and a stress agent, if no contraindications are present. The gadolinium based contrast agent to be used in this study is either Gadavist (up to 0.2 mL/kg body weight (0.2 mmol/kg) or MultiHance (0.2 mmol/kg) The IV stress agent is regadenoson (0.4mg/5ml bolus) or adenosine (dosage based on subject's weight and is set at 140mcg/kg/min
  Other Names: Myocardial Perfusion imaging; Myocardial Perfusion CMR; Magnetic Resonance Imaging; First Pass Myocardial Perfusion Imaging
Drug: Contrast — The intravenous gadolinium based contrast agent to be used in this study is either Gadavist (up to 0.2 mL/kg body weight (0.2 mmol/kg) or MultiHance (0.2 mmol/kg)
  Other Names: contrast media; Gadavist; MultiHance
Drug: Pharmacologic Stress Agent — The stress agent administered intravenously is regadenoson (0.4mg/5ml bolus) or adenosine (dosage based on subject's weight and is set at 140mcg/kg/min
  Other Names: regadenoson; adenosine; stress agent

SUMMARY:
This study hopes to provide significant technical improvement in a Myocardial Blood Flow (MBF) cardiac magnetic resonance (CMR) quantification technique to address challenges and technical limitations for MBF CMR. By developing and validating novel techniques to improve first-pass perfusion (FPP) cardiac MR, we propose to increase diagnostic accuracy by minimizing false positives and false negatives, allow for better evaluation and accurate quantification of total ischemic burden and reduce image and motion-induced artifacts.

The broad, long-term objective of the proposed project is to improve the prognosis of patients with myocardial ischemia caused by coronary artery disease (CAD) or coronary microvascular dysfunction (CMD).

DETAILED DESCRIPTION:
All subjects will receive cardiac MRI scans to diagnose CAD or CMD. MR perfusion scans will be performed twice per subject: once at rest, and once after administration of a pharmacologic stress agent. There will be a >15 minute delay between the two scans. A gadolinium-based contrast agent will be administered during each scan to allow measurement of myocardial blood flow. Once myocardial blood flow is quantified, the measurements will be compared to previous reference measurements (when available) from PET myocardial perfusion imaging in the CAD patient cohort and coronary reactivity testing (CRT) in the CMD patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* 60 healthy male or female (18 or older) participants
* 110 male or female adults (18 or older) who have undergone clinical myocardial perfusion imaging at CSMC and been diagnosed with Coronary Disease (CAD).
* 50 female adults (21 or older) who have undergone coronary reactivity testing at CSMC and been diagnosed with coronary microvascular disease (CMD).

Exclusion Criteria:

* MR imaging is contraindicated in persons with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers, neurostimulators, and infusion pumps.
* Persons with ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial, aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged.
* Patients who are pregnant, nursing, implanted with non MR-compatible intrauterine devices (IUD's)
* Persons unable to tolerate MRI imaging secondary to an inability to lie supine or severe claustrophobia.
* Persons who are non-compliant with visit instructions, including inability to lie still, hold breath or follow procedure instructions
* Persons whose renal function test does not meet CSMC standard of care MRI contrast protocol requirements (GFR <45ml/min).
* Persons with stated allergy to animal dander
* acute coronary syndrome or acute myocardial infarction or ongoing myocardial ischemia or ECG evidence of ongoing ischemia;
* patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support or prior/planned PCI or CABG;
* non-ischemic cardiomyopathy or more than moderate valvular disease;
* contraindication to stress agent (adenosine) including asthma or prior adverse reaction to adenosine
* contraindications for gadolinium contrast;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — CMD cohort will enroll female participants only.
Study Population: * 60 healthy male or female (18 or older) participants
  * 110 male or female adults (18 or older) who have undergone clinical myocardial perfusion imaging at CSMC and been diagnosed with Coronary Disease (CAD).
  * 50 female adults (21 or older) who have undergone coronary reactivity testing at CSMC and been diagnosed with coronary microvascular disease (CMD).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
CAD findings by MRI | Day One
  Accuracy (sensitivity and specificity) of MRI-based diagnosis of coronary artery disease (CAD) as compared to PET.
CMD findings by MRI | Day One
  Accuracy (sensitivity and specificity) of MRI-based diagnosis of coronary microvascular dysfunction (CMD), as compared to CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyang Fan, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No